CLINICAL TRIAL: NCT05317416
Title: A RANDOMIZED, 2-ARM, PHASE 3 STUDY OF ELRANATAMAB (PF-06863135) VERSUS LENALIDOMIDE IN PATIENTS WITH NEWLY DIAGNOSED MULTIPLE MYELOMA AFTER UNDERGOING AUTOLOGOUS STEM-CELL TRANSPLANTATION
Brief Title: Study With Elranatamab Versus Lenalidomide in Patients With Newly Diagnosed Multiple Myeloma After Transplant
Acronym: MagnetisMM-7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071007; MagnetisMM-7 (Other: Alias Study Number); 2023-508897-27-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: BCMA; Multiple Myeloma; Newly diagnosed; Elranatamab; Targeted T-cell; MagnetisMM; MM7; Phase 3; B-cell Maturation Antigen; monoclonal antibody; Stem cell transplant; Autologous stem cell transplant (ASCT); Hematologic disease; Minimum residual disease; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma; Hematologic Diseases | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A - Part 1 (Experimental): Elranatamab
  Interventions: Drug: Elranatamab
- Arm B - Part 1 (Active Comparator): Lenalidomide
  Interventions: Drug: Lenalidomide
- Arm B - Part 2 (Active Comparator): Lenalidomide
  Interventions: Drug: Lenalidomide
- Arm C - Part 2 (Experimental): Elranatamab
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Arms: Arm A - Part 1
Drug: Lenalidomide — Immunomodulatory drug
  Arms: Arm B - Part 1
Drug: Lenalidomide — Immunomodulatory drug
  Arms: Arm B - Part 2
Drug: Elranatamab — BCMA-CD3 bispecific antibody
  Arms: Arm C - Part 2

SUMMARY:
The purpose of this study is to evaluate whether elranatamab monotherapy can provide clinical benefit compared to lenalidomide monotherapy (control) in participants with newly diagnosed multiple myeloma after undergoing autologous stem cell transplant. In Part 1 and Part 2 of the study, participants in the study will either receive elranatamab (arm A and C) as an injection under the skin at the study clinic or lenalidomide orally once daily at home (arm B). Participation in the study will be approximately five years

DETAILED DESCRIPTION:
Elranatamab is a bispecific antibody: binding of elranatamab to CD3-expressing T-cells and BCMA-expressing multiple myeloma cells causes targeted T-cell-mediated cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM as defined according to IMWG criteria (Rajkumar, 2014) with measurable disease at diagnosis
* Part 1 patients must be MRD positive, Part 2 patients can be MRD negative or MRD positive
* History of induction therapy for newly diagnosed MM, followed by high dose therapy and autologous stem cell transplant. Randomization must occur within 120 days from the stem cell transplant. For participants who receive consolidation therapy after ASCT, randomization must occur within 60 days of consolidation and within 7 months from ASCT.
* Partial Response or better according to IMWG criteria at the time of randomization
* Must have an archival bone marrow aspirate sample(s) to identify the dominant malignant (index) clone by central laboratory NGS test (ClonoSEQ assay) that is used to track MRD status. This sample should preferably be collected before induction treatment (eg, at diagnosis) or before transplant.
* ECOG performance status ≤1
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤ 1
* Not pregnant and willing to use contraception

Exclusion Criteria:

* Plasma cell leukemia
* Amyloidosis, Waldenström's macroglobulinemia
* POEMS syndrome
* Known active CNS involvement or clinical signs of myelomatous meningeal involvement
* Previous MM maintenance treatment
* Prior treatment with BCMA targeted therapy
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) HBV, HCV, and known HIV or AIDS-related illness
* Previous administration with an investigational drug or vaccine within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2027-08-04 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease negativity rate | 12 months after randomization
  Minimal Residual Disease negativity rate per IMWG criteria as assessed via Next Generation Sequencing
Progression Free Survival | Assessed for up to approximately 5 years
  Progression Free Survival assessed by Blinded Independent Central review per IMWG response criteria

SECONDARY OUTCOMES:
Overall Survival | Assessed for up to approximately 5 years
  Defined as the time from randomization until death due to any cause
Sustained MRD negative rate | 24 months after randomization
  Sustained Minimal Residual Disease negative rate per IMWG criteria as assessed via Next Generation Sequencing
Progression Free Survival | Assessed for up to approximately 5 years
  Progression Free Survival by investigator per IMWG response criteria
Overall minimal residual disease negative rate | Assessed for up to approximately 5 years
  Minimal residual disease negative rate per IMWG criteria
Duration of minimal residual disease negativity | Assessed for up to approximately 5 years
  Minimal residual disease negativity per IMWG criteria
Sustained minimal residual disease negativity rate | Assessed for up to approximately 5 years
  Minimal residual disease negativity per IMWG criteria that has lasted a minimum of 12 months
Complete response rate | Assessed for up to approximately 5 years
  Complete response rate by blinded independent central review and by investigator per IMWG criteria
Duration of complete response | Assessed for up to approximately 5 years
  Duration of complete response by blinded independent central review and by investigator per IMWG criteria
Frequency of adverse events | Up to 90 days after last dose
  Adverse event as characterized by type, frequency, severity per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5, seriousness and relationship to the study intervention
Severity of Cytokine Release Syndrome and Immune effector Cell Associated Neurotoxicity syndrome | Assessed for up to approximately 5 years
  Cytokine Release Syndrome and Immune effector Cell Associated Neurotoxicity syndrome severity assessed per ASH-ASTCT criteria
Frequency of laboratory abnormalities | Assessed for up to approximately 5 years
Pre-dose concentrations of elranatamab | Assessed for up to approximately 5 years
  Pharmacokinetics of elranatamab (trough concentrations of elranatamab)
Post-dose concentrations of elranatamab | Assessed for up to approximately 5 years
  Pharmacokinetics of elranatamab (Post-dose serum concentrations of elranatamab)"
Incidence and titers of Anti-Drug Antibody and Neutralizing Antibody against elranatamab | Assessed for up to approximately 5 years
  Immunogenicity of elranatamab
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 | Assessed for up to approximately 5 years
  Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on symptom scales/items represent a greater presence of symptoms
Health-related quality of life by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Myeloma 20 | Assessed for up to approximately 5 years
  Higher scores on the functioning subscales (body image, future perspective) represent higher levels of functioning, whereas higher scores on the symptom subscales (disease symptoms, side effects) represent a greater presence of symptoms
Progression Free Survival 2 | Assessed for up to approximately 5 years
  Progression Free Survival to the date of second objective disease progression by investigator per IMWG response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (217):
- United States (24):
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner Gateway Medical Pavilion, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - Santa Monica UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Loyola University Chicago, Maywood, Illinois
  - Ascentist Doctor Hospital, Leawood, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - American Oncology Partners, P.A. Dba MidAmerica Cancer Care, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - WMCHealth Advanced Physician Services, Hawthorne, New York
  - Westchester Medical Center, Valhalla, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Arthur G.H. Bing, MD, Cancer Center, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Shoalhaven District Memorial Hospital, Nowra, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - QScan Radiology Clinics, Clayfield, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Epworth Healthcare, East Melbourne, Victoria
  - Precision Haematology, East Melbourne, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Slade Pharmacy, Richmond
- Austria (3):
  - Medizinische Universität Wien, Vienna, Vienna
  - Medizinische Universität Wien, Vienna
  - Hanusch-Krankenhaus, Vienna
- Belgium (7):
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi, Yvoir, Namur
  - UZ Gent, Ghent, Oost-vlaanderen
  - ZNA Middelheim, Antwerp
  - Zna Cadix, Antwerp
  - UZ Brussel, Brussels
- Brazil (16):
  - Instituto D'Or de Pesquisa e Ensino (IDOR) - Filial Salvador, Salvador, Estado de Bahia
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (USP), Ribeirão Preto, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo, São Paulo, São Paulo
  - Clínica Médica São Germano LTDA, SP, São Paulo
  - Fundação Doutor Amaral Carvalho, Jaú
  - Américas Medical City, Rio de Janeiro
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro
  - ESHO Empresa de Serviços Hospitalares S.A/ Hospital Samaritano de Higienópolis, São Paulo
  - HU UNIFESP / SPDM - Hospital São Paulo, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Hospital Japonês Santa Cruz, São Paulo
  - Clínica Médica São Germano S/S Ltda, São Paulo
- Canada (9):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Windsor Regional Hospital Cancer Program, Windsor, Ontario
  - Centre Integre Universitaire de la Santé et de Services Sociaux de l'Est-de-l'ile-de-Montreal,, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal (CIUSSS NÎ, Montreal, Quebec
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (5):
  - Fakultní nemocnice Brno Bohunice, Brno, Brno-město
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (3):
  - Oulun yliopistollinen sairaala, Oulu, North Ostrobothnia
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Uusimaa
- France (9):
  - Institut Universitaire du Cancer Toulouse - Oncopole - CHU de TOULOUSE, Toulouse, Haute-garonne
  - Pitie Salpetriere University Hospital, Paris, ORNE
  - Gustave Roussy, Villejuif, Val-de-marne
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Chu Grenoble Alpes, La Tronche
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Hôpital Saint Antoine, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau, Tours
- Germany (8):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Klinikum Chemnitz gGMbH, Chemnitz
  - Universitätsklinikum Essen, Essen
  - Klinikum rechts der Isar der Technischen Universität München, München
- Greece (3):
  - Alexandra General Hospital of Athens, Athens, Attikí
  - Theageneio Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - University Hospital of Ioannina, Ioannina, Ípeiros
- Hungary (5):
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Semmelweis University, Budapest
  - Dél-Pesti Centrumkórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Jósa András Oktatókórház, Nyíregyháza
- India (6):
  - Artemis hospital, Gurugram, Haryana
  - Medanta-The Medicity, Gurugram, Haryana
  - Fortis Memorial Research Institute, Gurugram, Haryana
  - Himalayan Institute Hospital Trust University, Dehradun, Uttarakhand
  - Tata Medical Center, Kolkata, West Bengal
  - Rajiv Gandhi Cancer Institute And Research Centre, Delhi
- Israel (9):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Hadassah Mount Scopus Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Soroka Medical Center, Beersheba, Southern District
  - Tel-Aviv Sourasky Medical Center Dana-Dwek Children's Hospital, Tel Aviv, TELL ABĪB
  - Shaare Zedek Medical Center, Jerusalem
- Italy (8):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Policlinico "G. Rodolico", Catania, Sicily
  - Azienda Ospedaliero Universitaria Senese, Siena, Tuscany
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - AOU Policlinico Umberto I, Roma
- Japan (16):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Iwate Medical University Hospital, Yahaba-cho, Iwate
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Japanese Red Cross Medical Center, Tokyo
- Netherlands (3):
  - HagaZiekenhuis, The Hague, South Holland
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Isala, Zwolle
- Norway (2):
  - Oslo Universitetssykehus Ullevål, Oslo
  - Stavanger Universitetssykehus, Stavanger
- Poland (7):
  - Centrum Medyczne Pratia Poznań, Skórzewo, Greater Poland Voivodeship
  - Pratia Onkologia Katowice, Katowice, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne,, Gdansk
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Uniwersyteckie Centrum Kliniczne WUM Centralny Szpital Kliniczny, Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- South Korea (10):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - Chonnam National University Hwasun Hospital, Hwasun Gun, Jeonranamdo
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital(Seoul St. Mary's Hospital), Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University, Daegu, Taegu-kwangyǒkshi
  - Kyungpook National University Hospital, Junggu, Taegu-kwangyǒkshi
- Spain (19):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet Del Llobregat, Barcelona [barcelona]
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona [barcelona]
  - Institut Catala d' Oncologia. Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Madrid, Madrid, Comunidad de
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital San Pedro de Alcántara, Cáceres
  - Institut Catala Oncologia - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (6):
  - Helsingborgs Lasarett, Helsingborg, Skåne LÄN [se-12]
  - Karolinska Universitetssjukhuset Huddinge, Stockholm, Stockholms LÄN [se-01]
  - Södra Älvsborgs Sjukhus Borås, Borås, Västra Götalands LÄN [se-14]
  - Falu Lasarett, Falun
  - Universitetssjukhuset Örebro, Örebro, Örebro LÄN [se-18]
  - Universitetssjukhuset i Linköping, Linköping, Östergötlands LÄN [se-05]
- Switzerland (5):
  - CHUV (centre hospitalier universitaire vaudois), Lausanne, Canton of Vaud
  - UniversitätsSpital Zürich, Zurich, Zürich (DE)
  - Kantonsspital Baden, Baden
  - Inselspital Bern, Bern
  - Kantonsspital Winterthur, Winterthur
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Medipol Mega Universite Hastanesi, Istanbul, İ̇stanbul
  - Sisli Florence Nightingale Hastanesi, Istanbul, İ̇stanbul
  - Ege Universitesi Hastanesi, Izmir, İ̇zmir
  - Dokuz Eylul Universitesi Hastanesi, Izmir, İ̇zmir
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Aydın Adnan Menderes Universitesi Hastanesi, Aydin
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri, Kayseri
  - Özel Anadolu Sağlık Merkezi, Kocaeli
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Queen Elizabeth Hospital Birmingham, Birmingham, England
  - Belfast City Hospital, Belfast
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Berkshire Hospital, Reading
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071007